CLINICAL TRIAL: NCT07154017
Title: Efficacy of Combining Movement Representation Techniques to Active Neural Mobilization in the Mechanosensitivity of the Median Nerve: A Pilot Study, Single-blind,Randomized, Crossover.
Brief Title: Efficacy of Combining Movement Representation Techniques to Active Neural Mobilization in the Mechanosensitivity of the Median Nerve in Asymptomatic Volunteers.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Maximiliano Venosta, Physioterapist, University of Gran Rosario
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 886/2024
Record Dates: First submitted 2025-08-18; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Median Nerve
Keywords: Movement Representation Techniques; Neural Mobilization; Mechanosensitivity

STUDY DESIGN:
Intervention Model Description: A Pilot Study, Single-blind,Randomized, Crossover.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Evaluators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of Movement Representation Techniques with Neural Mobilization Exercises (experimental) (Experimental): Combination of Movement Representation Techniques (Action observation, Motor imagery and Mirror therapy) with Neural Mobilization Exercises (Active neural mobilization of Median nerve)
  Interventions: Other: Combination of Movement Representation Techniques with neural mobilization exercises
- Neural Mobilization Excercises (control) (Active Comparator): Neural Mobilization Exercises (Active neural mobilization of Median nerve)
  Interventions: Other: Neural mobilization exercises

INTERVENTIONS:
Other: Combination of Movement Representation Techniques with neural mobilization exercises — The experimental intervention will be an exposition of movement representation techniques in an established sequential order, consisting of action observation, implicit/explicit motor imagery and visual feedback with a mirror in combination with neural mobilization exercises.
  Arms: Combination of Movement Representation Techniques with Neural Mobilization Exercises (experimental)
Other: Neural mobilization exercises — The control intervention will consist in three series of active neural mobilization exercises
  Other Names: Neurodinamics excercises
  Arms: Neural Mobilization Excercises (control)

SUMMARY:
The objective of this study will be to determine whether the combination of movement imaging techniques with neural mobilization (NM) exercises works to modify median nerve sensitivity to mechanical stimuli. Movement Representation Techniques (MRTs) are defined as therapeutic or training systems that neurophysiologically evoke a perceptual-cognitive representation of movement. They can be combined with the execution of actual movement or with afferent sensory stimulation (motor command). There is evidence demonstrating positive results in pain reduction and improved range of motion using MRTs alone.

The study will be evaluated in 10 randomly selected asymptomatic volunteers, considering the following variables: pressure pain threshold, elbow extensor range of motion, and sensory responses before and after the intervention, in both the experimental and control groups. The period between interventions will be 72 hours.

DETAILED DESCRIPTION:
The objective of this pilot study will be to determine the efficacy of combining movement representation techniques with neural mobilization (NM) exercises on median nerve mechanosensitivity. Movement representation techniques (MRTs) are defined as therapeutic or training systems that neurophysiologically evoke a perceptual-cognitive representation of movement through imagery or observation of motor actions. They can be combined with actual movement execution or with afferent sensory stimulation (motor command). There is evidence demonstrating positive results in pain reduction and range of motion gains using MRTs alone.

The study will be designed as a randomized, single-blind, crossover pilot clinical trial. In this study, 10 asymptomatic volunteers will be randomly selected and measured in the following variables: pressure pain threshold (PPT), elbow extensor range of motion (EROM), and the spatiotemporal distribution of pre- and post-intervention sensory responses in both the experimental group (RMM + MN) and the control group (MN). The washout period between interventions will be 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic volunteers of both sexes
* aged 18 to 45
* with no symptoms or history of disease in the cervical region, shoulder girdle, or upper limb.

Exclusion Criteria:

* history of surgery or trauma to the cervical spine, shoulder girdle, or upper limb;
* nonspecific shoulder pain;
* presenting symptoms of chronic pain in any region of the body;
* aphantasia (inability to create mental images);
* hypermobility;
* history of cancer or active disease;
* current infection;
* rheumatological disease;
* neurological and/or psychiatric disorders;
* altered sensation;
* current pregnancy;
* consumption of centrally acting medications;
* undergoing physiotherapy treatment in the last month;
* inability to understand the informed consent document;
* previous experience with median nerve provocation testing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Elbow Extensor Range of Motion | Pre- and post-interventions with a 72-hour washout period, for both control and experimental.
  The elbow extension movement will be measured during the median nerve provocation test, through digital inclinometry of both the dominant and non-dominant arm by an experienced Physiotherapist.
Pressure Pain Threshold | Pre and post interventions, both control and experimentalPre- and post-interventions with a 72-hour washout period, for both control and experimental.
  Pressure pain thresholds (PPTs) will be performed at two sites, the dominant and non-dominant side, in asymptomatic participants: 1) the upper trapezius muscle, and 2) the proximal third of the forearm. A pressure algometer will be used. The device has a rod at one end with a 1 cm2 flat, circular rubber tip. Pressure will be applied progressively in a perpendicular direction at a rate of 0.5 kgf/cm2 per second to the assessment sites. Volunteers will be asked to verbally report the moment they feel the pressure exerted with the pressure algometer begin to change to a sensation of pain (first painful sensation). At that moment, the evaluator will stop applying pressure and a value will be obtained. Three measurements will be taken at each site, 30 seconds apart. The PPT will be determined as the arithmetic mean of the three measurements.
Spatiotemporal distribution of sensory responses | Pre- and post-interventions with a 72-hour washout period, for both control and experimental.
  Humanoid software (University Center of Assistance, Teaching and Investigation, CUADI, Argentina) will be used to evaluate the spatiotemporal distribution of pain intensity and/or perceived sensations. To mark the sensations that subject feel during the arm stretch test. To do this, the subjects will mark the area on the touchscreen where they perceive tension or stretching. The sensations will be representated by different colours: yellow is used for mild sensations, orange for moderate sensations, and red for intense sensations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gran Rosario, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Yes, the statistical analysis and consent form
Supporting Information: SAP, ICF
Time Frame: From first date of publication of journal article.
Access Criteria: IPD will be provided upon request.

REFERENCES:
- [Result] Matesanz-Garcia L, Caceres-Pajuelo JE, Cuenca-Martinez F, La Touche R, Goicoechea-Garcia C, Fernandez-Carnero J. Effects of neural mobilizations through movement representation techniques for the improvement of neural mechanosensitivity of the median nerve region: a randomized controlled trial. Somatosens Mot Res. 2021 Dec;38(4):267-276. doi: 10.1080/08990220.2021.1964463. Epub 2021 Aug 17. PMID 34404324